CLINICAL TRIAL: NCT04704869
Title: A Multi-center, Randomized, Controlled Trial Evaluating the Effects of Early High-Dose Cryoprecipitate in Adult Patients With Major Trauma Hemorrhage Requiring Major Hemorrhage Protocol (MHP) Activation
Brief Title: Early Use of Cryoprecipitate With Major Hemorrhage Protocol (MHP) Activation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bryan Cotton (Other)
Collaborators: Queen Mary University of London (Other); NHS Blood and Transplant (Other Government)
Responsible Party: Sponsor-Investigator, Bryan Cotton, Professor of Surgery, The University of Texas Health Science Center, Houston
Organization: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-19-0272; ISRCTN14998314 (Registry Identifier: International Standard Randomised Controlled Trial Number)
Record Dates: First submitted 2021-01-06; First posted 2021-01-12 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries | interventions — cryoprecipitate coagulum; Erythrocyte Count; Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) (Experimental): Cryoprecipitate will be given in addition to the standard of care massive transfusion protocol products, which include red blood cells, plasma, platelets and whole blood. The Cryoprecipitate will be given with 90 minutes of emergency department arrival. Cryoprecipitate dose will be 3 pools (equivalent to 15 single units).
  Interventions: Biological: Cryoprecipitate; Biological: Red Blood Cells; Biological: Plasma; Biological: Platelets; Biological: Whole Blood
- Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) (Active Comparator): Only standard of care massive transfusion protocol products will be given, including red blood cells, plasma, platelets, and whole blood.
  Interventions: Biological: Red Blood Cells; Biological: Plasma; Biological: Platelets; Biological: Whole Blood

INTERVENTIONS:
Biological: Cryoprecipitate — Cryoprecipitate is a blood product high in fibrinogen. The Cryoprecipitate will be given with 90 minutes of emergency department arrival. Cryoprecipitate dose will be 3 pools (equivalent to 15 single units).
  Arms: Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Biological: Red Blood Cells — RBCs are utilized as part of the Massive Transfusion protocol for hemorrhage control.
  Other Names: RBCs
Biological: Plasma — Plasma is utilized as part of the Massive Transfusion protocol for hemorrhage control.
Biological: Platelets — Platelets are utilized as part of the Massive Transfusion protocol for hemorrhage control.
Biological: Whole Blood — Whole Blood is utilized as part of the Massive Transfusion protocol for hemorrhage control.

SUMMARY:
The purpose of this trial is to compare standard of care (SOC) massive transfusion protocol to SOC massive transfusion protocol plus early use of cryoprecipitate (within 90 minutes of emergency department arrival).

ELIGIBILITY:
Inclusion Criteria:

* The patient is judged to be an adult (according to local practice, e.g. 16 years or older in UK) and has sustained severe traumatic injury. In the event the age is unknown, estimated body weight ≥50 kg.
* The patient is deemed by the attending clinician to have on-going active hemorrhage AND REQUIRES Activation of the local major hemorrhage protocol for management of severe blood loss AND HAS STARTED or HAS RECEIVED at least one unit of any blood component

Exclusion Criteria:

* The patient has been transferred from another hospital
* The trauma team leader deems the injuries incompatible with life
* More than 3 hours have elapsed from the time of injury
* Prisoner (as defined as someone admitted from a correctional facility)
* Known "Do Not Resuscitate" orders
* Enrolled in a concurrent ongoing interventional, randomized clinical trial
* Patients who wear "opt out" bracelet for study
* Obvious pregnancy
* Severely burned

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1604 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan A Cotton, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (25):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States
- United Kingdom (24):
  - Queen Elizabeth Hospital, Birmingham
  - Royal Sussex County Hospital, Brighton
  - Southmead Hospital, Bristol
  - Addenbrooke's Hospital, Cambridge
  - University Hospital of Wales, Cardiff
  - University Hospital of Coventry and Warwickshire, Coventry
  - Hull Royal Infirmary, Hull
  - Leeds General Infirmary, Leeds
  - University Hospital Aintree, Liverpool
  - Royal London Hospital, London
  - King's College Hospital, London
  - St. George's Hospital, London
  - St. Mary's Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Salford Royal Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Queens Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Preston Hospital, Preston
  - Northern General Hospital, Sheffield
  - University Hospital Southampton, Southampton
  - University Hospital of North Staffordshire, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davenport R, Curry N, Fox EE, Thomas H, Lucas J, Evans A, Shanmugaranjan S, Sharma R, Deary A, Edwards A, Green L, Wade CE, Benger JR, Cotton BA, Stanworth SJ, Brohi K; CRYOSTAT-2 Principal Investigators. Early and Empirical High-Dose Cryoprecipitate for Hemorrhage After Traumatic Injury: The CRYOSTAT-2 Randomized Clinical Trial. JAMA. 2023 Nov 21;330(19):1882-1891. doi: 10.1001/jama.2023.21019. PMID 37824155

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Started | 805 | 799
Completed 28-day Follow up | 771 | 760
Completed | 771 | 760
Not Completed | 34 | 39

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Total
Number analyzed (Participants) | 799 | 805 | 1604
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age data were not be collected for 9 in the Massive Transfusion Protocol arm and for 14 in the Early Cryoprecipitate plus Massive Transfusion Protocol arm.
  years
    number analyzed (Participants) | 785 | 796 | 1581
    (all) | 38 [25 to 55] | 40 [26 to 55] | 39 [26 to 55]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex data were not be collected for 9 in the Massive Transfusion Protocol arm and for 14 in the Early Cryoprecipitate plus Massive Transfusion Protocol arm.
  Participants
    number analyzed (Participants) | 785 | 796 | 1581
    Female | 167 | 163 | 330
    Male | 618 | 633 | 1251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity data were only collected from 48 US participants.
  Participants
    number analyzed (Participants) | 24 | 24 | 48
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 16 | 14 | 30
    Unknown or Not Reported | 8 | 9 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race data were only collected from 48 US participants.
  Participants
    Race: number analyzed (Participants) | 24 | 24 | 48
    Race: Black | 10 | 6 | 16
    Race: White | 5 | 8 | 13
    Race: Other | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 24 | 25 | 48
  United Kingdom | 775 | 780 | 1555
Time from injury to ED arrival [Median (Inter-Quartile Range); unit: minutes] | 75 [55 to 99] | 77 [55 to 100] | 76 [55 to 100]
Number of Participants who arrived at the Emergency Department with a blunt injury [Count of Participants; unit: Participants] — Population: Number of participants who arrived in the Emergency Department with a blunt injury data were not be collected for 9 in the Massive Transfusion Protocol arm and for 14 in the Early Cryoprecipitate plus Massive Transfusion Protocol arm.
  Participants
    number analyzed (Participants) | 785 | 796 | 1581
    (all) | 495 | 519 | 1014
Number of Participants who arrived to the Emergency Department in cardiac arrest [Count of Participants; unit: Participants] — Population: Number of participants who arrived to the Emergency Department in cardiac arrest were not be collected for 70 in the Massive Transfusion Protocol arm and for 82 in the Early Cryoprecipitate plus Massive Transfusion Protocol arm.
  Participants
    number analyzed (Participants) | 717 | 735 | 1452
    (all) | 12 | 17 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mortality From Any Cause
Description: Mortality from any cause
Time Frame: 28 days after emergency department (ED) admission
Population: Vital status was not available from any source for 34 in the Massive Transfusion Protocol arm and 39 in the Early Cryoprecipitate plus Massive Transfusion Protocol arm. Data presented are from an intention to treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 771 | 760
Participants | 201 | 192
Statistical Analysis 1: Comparison: Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) vs Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood); Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.81 to 1.17]

2. Secondary Outcome: All Cause Mortality at 6 Hours
Description: Mortality from any cause
Time Frame: 6 hours after ED admission
Population: Data were not collected for 15 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected for 10 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 784 | 795
Participants | 56 | 68

3. Secondary Outcome: All Cause Mortality at 24 Hours
Description: Mortality from any cause
Time Frame: 24 hours after ED admission
Population: Data were not collected for 16 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected for 11 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm
Measure: Count of Participants; unit: Participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 783 | 794
Participants | 88 | 97

4. Secondary Outcome: All Cause Mortality at 6 Months
Description: Mortality from any cause. All cause mortality at 6 months is presented as a Kaplan-Meier estimated.
Time Frame: 6 months after ED admission
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 799 | 805
percentage of participants | 26.1 [23.2 to 29.4] | 27.3 [24.3 to 30.7]

5. Secondary Outcome: All Cause Mortality at 12 Months
Description: Mortality from any cause. All cause mortality at 6 months is presented as a Kaplan-Meier estimated.
Time Frame: 12 months after ED admission
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 799 | 805
percentage of participants | 26.6 [23.6 to 30.0] | 27.7 [24.6 to 31.1]

6. Secondary Outcome: Death From Bleeding at 6 Hours
Description: Death related to exsanguination
Time Frame: 6 hours after ED admission
Population: Data were not collected from 10 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 15 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 784 | 795
Participants | 32 | 35

7. Secondary Outcome: Death From Bleeding at 24 Hours
Description: Death related to exsanguination
Time Frame: 24 hours after ED admission
Population: Data were not collected from 11 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 16 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 783 | 794
Participants | 43 | 39

8. Secondary Outcome: Transfusion Requirements (Number of Units of Red Blood Cells (RBCs))
Description: Number of units of RBCs
Time Frame: from time of pre-hospital care to 24 hours after ED admission, an average of 30 hours
Population: Data were not collected from 108 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 104 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Median (Inter-Quartile Range); unit: Units
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 695 | 697
Units | 5 [3 to 9] | 5 [3 to 8]

9. Secondary Outcome: Transfusion Requirements (Number of Units of Plasma)
Description: Number of units of plasma
Time Frame: from time of pre-hospital care to 24 hours after ED admission, an average of 30 hours
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 695 | 697
units | 4 [2 to 8] | 4 [2 to 8]

10. Secondary Outcome: Transfusion Requirements (Number of Units of Platelets)
Description: Number of units of platelets
Time Frame: from time of pre-hospital care to 24 hours after ED admission, an average of 30 hours
Population: Data were not collected from 110 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 104 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Median (Inter-Quartile Range); unit: Units
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 695 | 695
Units | 0 [0 to 1] | 0 [0 to 1]

11. Secondary Outcome: Transfusion Requirements (Number of Units of Cryoprecipitate)
Description: Number of units of cryoprecipitate
Time Frame: from time of pre-hospital care to 24 hours after ED admission, an average of 30 hours
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Units
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 695 | 695
Units | 3 [3 to 3] | 0 [0 to 2]

12. Secondary Outcome: Destination of Participant at Time of Discharge From Hospital
Description: Destination of participant at time of discharge from hospital
Time Frame: at the time of discharge from hospital, about 11-27 days after admission
Population: Data were not collected from 431 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 424 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 375 | 374
Participants
  Home | 280 | 278
  Nursing home/rehabilitation facility | 9 | 8
  Other hospital | 63 | 72
  Other | 23 | 16

13. Secondary Outcome: Quality of Life as Assessed by EuroQol-5 Dimension-5 Level (EQ5D-5L)
Description: The 5-level EQ-5D version (EQ-5D-5L) score range was -0.148 (worst health state) to 0.949 (best health state). A higher score indicating a better health state.
Time Frame: Day of hospital discharge or 28 days after ED admission (whichever comes first)
Population: Data were not collected from 458 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 475 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 324 | 347
score on a scale | 0.51 [0.26 to 0.72] | 0.50 [0.20 to 0.73]

14. Secondary Outcome: Quality of Life as Assessed by the Glasgow Outcome Score
Description: The Glasgow Outcome Score ranges from 1 to 5, with a higher score indicating a better outcome:
  1. Death - Severe injury or death without recovery of consciousness
  2. Persistent vegetative state - Severe damage with prolonged state of unresponsiveness and a lack of higher mental functions
  3. Severe disability - Severe injury with permanent need for help with daily living
  4. Moderate disability - No need for assistance in everyday life, employment is possible but may require special equipment
  5. Low disability - Light damage with minor neurological and psychological deficits
Time Frame: Day of hospital discharge or 28 days after ED admission (whichever comes first)
Population: Data were not collected from 93 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 94 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 705 | 712
Participants
  Low disability | 226 | 221
  Moderate disability | 129 | 129
  Severe disability | 155 | 153
  Persistent vegetative state | 21 | 27
  Death | 174 | 182

15. Secondary Outcome: Quality of Life as Assessed by EuroQol-5 Dimension-5 Level (EQ5D-5L)
Description: as for outcome 13
Time Frame: 6 months after ED admission
Population: Data were not collected from 350 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 331 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 468 | 455
score on a scale | 0.76 [0.63 to 0.93] | 0.66 [0.36 to 0.78]

16. Secondary Outcome: Quality of Life as Assessed by the Glasgow Outcome Score
Description: as for outcome 14
Time Frame: 6 months after ED admission
Population: Data for this outcome measure were not collected because the survey was not included on the 6-month follow-up. As a result, no participants received the survey, and therefore, no participants were analyzed in either study arm.
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Hospital Resource Use as Assessed by Number of Ventilator Days
Description: Number of ventilator days during hospitalization
Time Frame: Day of hospital discharge or 28 days after ED admission (whichever comes first)
Population: Data were not collected from 34 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 36 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 763 | 771
days | 1 [0 to 6] | 1 [0 to 7]

18. Secondary Outcome: Hospital Resource Use as Assessed by Number of Intensive Care Unit (ICU) Days
Description: Number of ICU days during hospitalization
Time Frame: Day of hospital discharge or 28 days after ED admission (whichever comes first)
Population: as for outcome 17
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 763 | 771
days | 4 [1 to 12] | 4 [1 to 13]

19. Secondary Outcome: Hospital Resource Use as Assessed by Number of Hospital Days
Description: Total number of hospital days
Time Frame: Day of hospital discharge or 28 days after ED admission (whichever comes first)
Population: Data were not collected from 33 participants in the Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm. Data were not collected from 36 participants in the Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) arm.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
Number analyzed (Participants) | 763 | 772
days | 11 [3 to 27] | 11 [3 to 27]

ADVERSE EVENTS:
Time Frame: Day of hospital discharge or 28 days after ED admission (whichever comes first)
Description: 28-day vital status was not available from any source for 34 in the Massive Transfusion arm and 39 in the Early Cryoprecipitate + Massive Transfusion arm; therefore, all-Cause Mortality data could not be assessed for 34 in the Massive Transfusion arm and 39 in the Early Cryoprecipitate + Massive Transfusion arm.
Arm/Group | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood)
All-Cause Mortality (participants affected / at risk) | 201/771 | 192/760
Serious Adverse Events (participants affected / at risk) | 83/805 | 84/799
Other Adverse Events (participants affected / at risk) | 0/805 | 0/799
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) (N=805) | Early Cryoprecipitate + Massive Transfusion Protocol (RBCs, Plasma, Platelets, Whole Blood) (N=799)
Venous thromboembolism (Vascular disorders) | 57 (59) | 55 (58)
Arterial thrombotic event (Vascular disorders) | 26 (26) | 26 (27)
Serious transfusion related adverse event (General disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT04704869/Prot_SAP_000.pdf